CLINICAL TRIAL: NCT02415699
Title: Randomized Controlled Trial Comparing DC-CIK Immunotherapy Combined With Adjuvant Chemotherapy and Adjuvant Chemotherapy Alone in Stage III Colorectal Cancer.
Brief Title: DC-CIK Immunotherapy Plus Chemotherapy vs Chemotherapy Alone in the Adjuvant Treatment of Stage III Colorectal Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015045010
Record Dates: First submitted 2015-04-09; First posted 2015-04-14 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Oxaliplatin; Leucovorin

ARMS (2):
- DC-CIK Immunotherapy Plus Chemotherapy (Experimental): Stage III Colon Cancer patients after radical operation and adjuvant chemotherapy will receive 12 cycles of DC-CIK therapy in this group
  Interventions: Drug: Fluorouracil; Drug: Oxaliplatin; Drug: Leucovorin; Biological: DC-CIK
- Chemotherapy Alone (Active Comparator): Stage III Colon Cancer patients after radical operation and adjuvant chemotherapy alone.
  Interventions: Drug: Fluorouracil; Drug: Oxaliplatin; Drug: Leucovorin

INTERVENTIONS:
Drug: Fluorouracil
  Other Names: 5-FU
Drug: Oxaliplatin
Drug: Leucovorin
Biological: DC-CIK
  Arms: DC-CIK Immunotherapy Plus Chemotherapy

SUMMARY:
Stage III colorectal cancer constitutes more than half of the colorectal patients, and the prognosis does not improve much recently although varies of adjuvant drugs have been tried. DC-CIK immunotherapy has been proved to improve survival in cancer patients, but its role in stage III colorectal cancer patients stains unclear. The investigators study will focus on the efficacy and safety of DC-CIK immunotherapy plus chemotherapy in the adjuvant treatment of stage III colorectal cancer, compared with chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Stage III colon cancer
* Undergone complete resection of primary tumor
* Completed standard adjuvant chemotherapy
* ECOG performancer status 0-2
* Adequate hematologic, hepatic and renal functions

Exclusion Criteria:

* HIV positive or other Immunodeficiency disease
* Uncontrolled hypertension
* History of recent cancers in the past 5 years
* Patients with previous or concurrent malignancy or any anti-cancer therapy
* Patients who were allergic to platinum drugs or fluorouracil
* Pregnant patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 2 years

SECONDARY OUTCOMES:
Overall survival | 2 years
Side Effect | 6 month